CLINICAL TRIAL: NCT04640610
Title: Study of the Expression of Angiotensin-converting Enzyme 2 (ACE2), a Cell Membrane Receptor for SARS-CoV-2 and the TMPRSS2 Serine Protease in Tonsils and Adenoids of Children and Adults
Brief Title: Angiotensin-converting Enzyme 2 (ACE2) Expression in Tonsils and Adenoids
Acronym: ACE2-AVG
Status: Withdrawn | Type: Observational
Why Stopped: Abandonment of the study project
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201032
Record Dates: First submitted 2020-11-19; First posted 2020-11-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2021-06

CONDITIONS: Adenoidectomy; Tonsillectomy
Keywords: SARS-CoV-2; Angiotensin-converting enzyme 2 (ACE2); Transmembrane serine protease 2 (TMPRSS2); Tonsils; Adenoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tonsils and adenoids preserved by cryopreservation and fixed with formalin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adenoidectomy / tonsillectomy: Children and adults, without SARS-CoV-2 infection, in whom an adenoidectomy and/or tonsillectomy is performed for their care in the centers of the study.
  Interventions: Other: Storage of operating waste

INTERVENTIONS:
Other: Storage of operating waste — Storage of operating waste of adenoidectomy / tonsillectomy

SUMMARY:
The objective of the research is to study the expression of the ACE 2 receptor and the TMPRSS2 serine protease in the tonsils and adenoids of children and adults.

DETAILED DESCRIPTION:
The entry point for SARS-CoV-2 into the body is the nasal and pharyngeal mucosa. Angiotensin-converting enzyme 2 (ACE 2) was quickly identified as the functional receptor for SARS-CoV-2. Furthermore, the TMPRSS2 serine protease is required for the anchoring of the S protein in cell lines. In addition, the most commonly used screening test is a test for viral RNA by RT-PCR on a nasopharyngeal sample because the viral load is high.

The tonsils and adenoids could be a target organ of the virus. In order to study this hypothesis, the expression of ACE 2 and the serine protease TMPRSS2 will be sought in these tissues.

In addition, children, generally at high risk of severe viral respiratory infections (RSV, influenza), have milder symptoms than older patients with SARS-CoV-2 infection. The reason for this difference remains elusive. But one of the hypotheses formulated is that the level of expression of ACE 2 and / or TMPRSS2 may differ between adults and children, the viral load seeming to be correlated with the severity of the attack. In order to study this hypothesis, we will therefore compare the level of expression of ACE 2 in the tonsil tissue of children and adults.

ELIGIBILITY:
Inclusion Criteria:

* Children and adults, without SARS-CoV-2 infection, in whom an adenoidectomy and/or tonsillectomy is performed for their care in the hospitals of Assistance Publique-Hôpitaux de Paris participating in the study.
* Holders of parental authority of minor patients and adult patients not opposed to participation in the study.

Exclusion Criteria:

- N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults, without SARS-CoV-2 infection, in whom an adenoidectomy and/or tonsillectomy is performed for their care in the centers of the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Expression of ACE 2 receptor and TMPRSS2 serine protease | 9 months
  Measurement of expression of ACE 2 receptor and TMPRSS2 serine protease in tonsils and adenoids labeled by immunofluorescence.

SECONDARY OUTCOMES:
Location of ACE 2 receptor and TMPRSS2 serine protease | 9 months
  Location of ACE 2 receptor and TMPRSS2 serine protease in tonsils and adenoids labeled by immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Luscan, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Pierre-Louis Tharaux, MD, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (9):
- France (9):
  - Hôpital Mondor, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Lariboisière, Paris
  - Hôpital Armand Trousseau, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - HEGP, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Bichat, Paris
  - Hôpital Tenon, Paris

IPD SHARING:
Plan to Share IPD: No